CLINICAL TRIAL: NCT02887014
Title: Providing Specific Verbal Instructions Improves Bowel Preparation of Inpatients Undergoing Colonoscopy: a Multi-center Single Blinded Randomized Study
Brief Title: Specific Verbal vs. Usual Instructions for Inpatients Undergoing Colonoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Attikon Hospital (Other)
Collaborators: University Hospital, Ioannina (Other); University Hospital of Patras (Other); Larissa University Hospital (Other)
Responsible Party: Principal Investigator, ATHANASIOS SIOULAS, Dr, Attikon Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: INPATIENTS_VERBAL-001
Record Dates: First submitted 2016-08-15; First posted 2016-09-01 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Adequate Colonoscopy Preparation for Inpatients
Keywords: bowel preparation; colonoscopy; inpatients; cathartics

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Participants getting SPECIFIC VERBAL INSTRUCTIONS before starting bowel preparation (Group A).
  Interventions: Procedure: SPECIFIC VERBAL INSTRUCTIONS
- Group B (No Intervention): Participants getting ordinary instructions as usual in each of the participating centers (Group B).

INTERVENTIONS:
Procedure: SPECIFIC VERBAL INSTRUCTIONS — Participants will be randomized either to get detailed instructions verbally by the medico-paramedical staff of the participating centers (physicians or nurses) before starting bowel preparation (Group A) or to get ordinary instructions as usual in each of the participating centers (Group B). Instructions provided to Group A will include details about the procedure of bowel preparation, its potential side effects and the importance of the adequate preparation (Appendix)
  Arms: Group A

SUMMARY:
To study the impact of providing specific verbal instructions in inpatients (and/or their relatives) undergoing colonoscopy on the quality of bowel preparation.

DETAILED DESCRIPTION:
Introduction Adequate bowel preparation constitutes one of the most important endoscopy quality indicators: it is related with increased detection of pathologic findings, reduces the need for repeated colonoscopies and leads to burden lightening for both patients and endoscopy departments. Different factors have been related to inadequate preparation. Among them, inpatient status has been identified as a major independent risk factor.

It has been shown that providing outpatients with simple, but specific instructions regarding the importance and mode of adequate preparation - either through a leaflet, a sms or on the web - improves significantly the level of bowel cleanliness. However, data regarding the success of such an intervention in inpatients lack.

Aim To study the impact of providing specific verbal instructions in inpatients (and/or their relatives) undergoing colonoscopy on the quality of bowel preparation.

Patients - Methods Study Design This is a prospective, randomized, single-blinded study. Four Greek academic endoscopy departments will competitively enroll patients during a period of 6 months.

Randomization A central randomization list will be computer-assisted, created and sent to one collaborator of each center. Endoscopists will be blinded to participant's group.

300 patients will be randomized in 2 groups, in blocks of 10 with an analogy 1:1. They will also be stratified in a 60%-40% percentage depending on whether the patient is bedridden or not at the time of the examination

Statistical Analysis According to the literature similar interventions showed a gain of 20% in favor of the intervention. Statistical significance level α is defined 5% and the study is powered at the level of 80%. According to data from Hepatogastroenterology Unit of Attikon University General Hospital regarding the adequateness of bowel preparation of patients undergoing colonoscopy and with an expected 10% drop out, 300 patients are needed (including a 10% drop out) in order to succeed 18% improvement of the primary endpoint (from 66% for inpatients during 2015 to 84% for outpatients during the same period) favoring the intervention group. Interim analysis and sample size re-estimation will be undergone after data collection from 90 patients.

Both an intention to treat (ITT) and a per protocol (PP) analysis are planned. Data will be recorded in predefined CRFs.

ELIGIBILITY:
Inclusion Criteria:

* assignment of informed consent

Exclusion Criteria:

* inability to provide informed consent
* history of colectomy
* indication for rectosigmoidoscopy
* lack of knowledge of the Greek language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Increase in the number of examinations with adequate bowel preparation | At colonoscopy completion
  Bowel preparation will be considered adequate if overall BBPS≥6 and all segments achieving BBPS≥2.

SECONDARY OUTCOMES:
Overall BBPS score change | At colonoscopy completion
Segmental BBPS score changes | At colonoscopy completion
Total examination time, cecal intubation time and time needed to washout during the colonoscopy | At colonoscopy completion
Cecal intubation rate | At cecum intubation
Percentage of patients who received the whole amount of liquid preparation | Before colonoscopy start
Polyp and adenoma detection rate (overall and per segment) | Up to 4 weeks after patient's enrollment
Side effects related either to the preparation or the examination | Before colonoscopy start
  A questionnaire will be used as assessment method
Identification of potential additional risk factors for inadequate preparation | After colonoscopy completion
  Identification of potential additional risk factors for inadequate preparation (e.g. a bed status, performance status, autonomy level (measured by the Katz score) ΑSA Score, diabetes, use of tricyclic antidepressants, history of inadequate bowel preparation, chronic constipation, history of abdominal surgery other than colectomy, use of opioids, proposed predictive score. A questionnaire will be used.
Patient satisfaction from the bowel preparation using the visual analogue scale. | After colonoscopy completion

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Triantafyllou, Ass. Prof., Principal Investigator — Attikon Hospital
Locations (1):
- Hepatogastroenterology Unit, 2nd Department of Internal Medicine and Research Unit, Attikon University General Hospital, Athens, Greece

REFERENCES:
- [Background] Dik VK, Moons LM, Huyuk M, van der Schaar P, de Vos Tot Nederveen Cappel WH, Ter Borg PC, Meijssen MA, Ouwendijk RJ, Le Fevre DM, Stouten M, van der Galien O, Hiemstra TJ, Monkelbaan JF, van Oijen MG, Siersema PD; Colonoscopy Quality Initiative. Predicting inadequate bowel preparation for colonoscopy in participants receiving split-dose bowel preparation: development and validation of a prediction score. Gastrointest Endosc. 2015 Mar;81(3):665-72. doi: 10.1016/j.gie.2014.09.066. Epub 2015 Jan 17. PMID 25600879
- [Background] Ergen WF, Pasricha T, Hubbard FJ, Higginbotham T, Givens T, Slaughter JC, Obstein KL. Providing Hospitalized Patients With an Educational Booklet Increases the Quality of Colonoscopy Bowel Preparation. Clin Gastroenterol Hepatol. 2016 Jun;14(6):858-864. doi: 10.1016/j.cgh.2015.11.015. Epub 2015 Dec 8. PMID 26681487
- [Background] Guo X, Yang Z, Zhao L, Leung F, Luo H, Kang X, Li X, Jia H, Yang S, Tao Q, Pan Y, Guo X. Enhanced instructions improve the quality of bowel preparation for colonoscopy: a meta-analysis of randomized controlled trials. Gastrointest Endosc. 2017 Jan;85(1):90-97.e6. doi: 10.1016/j.gie.2016.05.012. Epub 2016 May 14. PMID 27189659
- [Background] Kumar A, Lin L, Bernheim O, Bagiella E, Jandorf L, Itzkowitz SH, Shah BJ. Effect of Functional Status on the Quality of Bowel Preparation in Elderly Patients Undergoing Screening and Surveillance Colonoscopy. Gut Liver. 2016 Jul 15;10(4):569-73. doi: 10.5009/gnl15230. PMID 27021501
- [Background] Lee YJ, Kim ES, Park KS, Cho KB, Jang BK, Chung WJ, Hwang JS. Education for Ward Nurses Influences the Quality of Inpatient's Bowel Preparation for Colonoscopy. Medicine (Baltimore). 2015 Aug;94(34):e1423. doi: 10.1097/MD.0000000000001423. PMID 26313794
- [Background] Rotondano G, Rispo A, Bottiglieri ME, De Luca L, Lamanda R, Orsini L, Bruzzese D, Galloro G; SIED Campania PISCoPO study group investigators; Romano M, Miranda A, Loguercio C, Esposito P, Nardone G, Compare D, Magno L, Ruggiero S, Imperatore N, De Palma GD, Gennarelli N, Cuomo R, Passananti V, Cirillo M, Cattaneo D, Bozzi RM, D'Angelo V, Marone P, Riccio E, De Nucci C, Monastra S, Caravelli G, Verde C, Di Giorgio P, Giannattasio F, Capece G, Taranto D, De Seta M, Spinosa G, De Stefano S, Familiari V, Cipolletta L, Bianco MA, Sansone S, Galasso G, De Colibus P, Romano M, Borgheresi P, Ricco G, Martorano M, Gravina AG, Marmo R, Rea M, Maurano A, Labianca O, Colantuoni E, Iuliano D, Trovato C, Fontana A, Pasquale L, Morante A, Perugini B, Scaglione G, Mauro B. Quality of bowel cleansing in hospitalized patients undergoing colonoscopy: A multicentre prospective regional study. Dig Liver Dis. 2015 Aug;47(8):669-74. doi: 10.1016/j.dld.2015.04.013. Epub 2015 Apr 25. PMID 26028360
- [Background] Srisarajivakul N, Chua D, Williams R, Leigh L, Ou A, Quarta G, Poles MA, Goodman A. How We Cleaned It Up: A Simple Method That Improved Our Practice's Bowel Prep. Am J Gastroenterol. 2016 Aug;111(8):1079-81. doi: 10.1038/ajg.2016.148. Epub 2016 Apr 26. No abstract available. PMID 27113117
- [Background] Yadlapati R, Johnston ER, Gregory DL, Ciolino JD, Cooper A, Keswani RN. Predictors of Inadequate Inpatient Colonoscopy Preparation and Its Association with Hospital Length of Stay and Costs. Dig Dis Sci. 2015 Nov;60(11):3482-90. doi: 10.1007/s10620-015-3761-2. Epub 2015 Jun 21. PMID 26093612